CLINICAL TRIAL: NCT05302219
Title: Plethysmography Curve Variability Depending on the Breath Cycle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Czech Technical University in Prague (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Plethysmography2022
Record Dates: First submitted 2022-03-16; First posted 2022-03-31 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Apnea; Circulatory; Change; Respiration
Keywords: pulse oximetry; photoplethysmography curve; breath cycle; apnea
MeSH Terms: conditions — Apnea; Respiratory Aspiration | interventions — Respiratory Rate; Tidal Volume; N(6)-2-(4-aminophenyl)ethyladenosine

STUDY DESIGN:
Intervention Model Description: All participants go through all assigned interventions in one study arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Measurement of plethysmography curve (Experimental): Calm measurement of plethysmography curve using pulse oximetry with simultaneous monitoring of the breath cycle. In this experimental arm, participants will vary their breath cycle (different respiratory rates and different tidal volumes).
  Interventions: Other: Respiratory rate; Other: Tidal volume; Other: Apnea

INTERVENTIONS:
Other: Respiratory rate — The participant alternates respiratory rates of 30, 15 and 7.5 breaths/min. Breathe each frequency for 2 minutes with a one-minute break.
Other: Tidal volume — The participant alternates tidal volumes of approx. 2, 1 and 0.5 litres. Breathe each tidal volume for 2 minutes with a one-minute break.
Other: Apnea — The participant simulates three apneic pauses lasting 1 minute with a two-minute break.

SUMMARY:
The aim of the study is to analyze the variability of plethysmography curve depending on the breath cycle (respiratory rate and tidal volume).

DETAILED DESCRIPTION:
The plethysmography curve measured by finger sensors using pulse oximetry shows the changes in blood volume at the measured site. The presence of respiratory information within the pulse oximeter signal is a well-documented phenomenon. However, previous studies have mainly focused on extracting the respiratory rate from the plethysmography curve. The aim of this study is to analyze the variability of plethysmography curve as a function of both respiratory rate and tidal volume. Furthermore, the aim is to analyze the possibilities of apneic pause detection from the plethysmography curve.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers/students from the Czech Technical University in Prague

Exclusion Criteria:

* any acute illness
* pregnancy
* severe cardiovascular conditions
* severe asthma or other severe respiratory conditions
* diabetes
* hypotension or hypertension

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Variability of plethysmography curve depending on the respiratory rate | 1 hour
  The effect of different respiratory rates (including apnea-zero respiratory rate) on the shape of the plethysmography curve will be evaluated.
Variability of plethysmography curve depending on the tidal volume | 1 hour
  The effect of different tidal volumes (including apnea-zero tidal volume) on the shape of the plethysmography curve will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Veronika Rafl Huttova, MSc, Principal Investigator — Czech Technical University in Prague; Jakub Rafl, PhD, Principal Investigator — Czech Technical University in Prague
Locations (1):
- Faculty of Biomedical Engineering, Czech Technical University in Prague, Kladno, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nilsson LM. Respiration signals from photoplethysmography. Anesth Analg. 2013 Oct;117(4):859-865. doi: 10.1213/ANE.0b013e31828098b2. Epub 2013 Feb 28. PMID 23449854